CLINICAL TRIAL: NCT04266756
Title: A Single-center, Open-label, Randomized, Formulation Screening, Two-cohort, Four-period, Crossover Study for Selexipag Sustained Release in Healthy Male Subjects
Brief Title: A Study of Selexipag in Healthy Male Participant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108709; 2019-004150-29 (EudraCT Number); 67896049PAH1001 (Other: Actelion)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Selexipag Matrix Tablets (Experimental): Participants will receive oral doses of selexipag matrix tablets based on release profiles (IR=immediate release, F=fast release, M=medium release and S=slow release) in treatment sequence 1 (IR+F+M+S), treatment sequence 2 (F+S+IR+M), treatment sequence 3 (M+ IR+ S+F) and treatment sequence 4 (S+M+F+IR) in periods 1, 2, 3, and 4, respectively under fasted condition. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Selexipag matrix tablet; Drug: Selexipag Immediate-release (IR) tablet
- Cohort 2: Selexipag Encapsulated Pellets (Experimental): Participants will receive oral doses of selexipag encapsulated) pellets based on release profiles (IR=immediate release, F=fast release, M=medium release and S=slow release) in treatment sequence 1 (IR+F+M+S), treatment sequence 2 (F+S+IR+M), treatment sequence 3 (M+ IR+ S+F) and treatment sequence 4 (S+M+F+IR) in periods 1, 2, 3, and 4, respectively under fasted condition. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Selexipag encapsulated pellets; Drug: Selexipag Immediate-release (IR) tablet

INTERVENTIONS:
Drug: Selexipag matrix tablet — Participants will receive single oral dose of Selexipag tablet(with fast, medium, and slow release profile) under fasted condition.
  Other Names: JNJ-67896049
  Arms: Cohort 1: Selexipag Matrix Tablets
Drug: Selexipag encapsulated pellets — Participants will receive single oral dose of Selexipag pellets (with fast, medium, and slow release profile) under fasted condition.
  Other Names: JNJ-67896049
  Arms: Cohort 2: Selexipag Encapsulated Pellets
Drug: Selexipag Immediate-release (IR) tablet — Participants will receive Selexipag immediate-release tablet orally under fasted condition.
  Other Names: JNJ-67896049

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) of selexipag and ACT-333679 following single oral administration of the matrix tablet and the encapsulated pellets of selexipag, each with 3 different release profiles, as compared to selexipag immediate release (IR) tablets in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participants may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must sign an informed consent form (ICF) indicating they understand the purpose of, and procedures required for, the study and is willing to participate in the study
* Body mass index (BMI; weight (kilogram [kg]/height^2 [meter {m}]^2) between 18.0 and 28.0 kilogram per square centimeter (kg/m^2) (inclusive), and body weight not less than 50.0 kg at screening
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 145 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening. If blood pressure is out of range, up to 2 repeated assessments within the screening period are permitted, last assessment being conclusive

Exclusion Criteria:

* Clinically significant abnormal values for hematology, biochemistry, or urinalysis at screening and on Day -1 of Treatment Period 1 as deemed appropriate by the investigator
* Known allergies, hypersensitivity, or intolerance to selexipag or its excipients
* Any contraindication included in the Summary of Product Characteristics (SmPC) of selexipag
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study treatments (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Previous history of stroke, fainting, collapse, syncope, orthostatic hypotension, vasovagal reactions, head injury

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Selexipag and ACT-333679 | Predose and 0 to 72 hours postdose
  The Cmax is the maximum observed analyte concentration.
Area Under Analyte Concentration From Time Zero to the Last Quantifiable Concentration (AUC [0-last]) of Selexipag and ACT-333679 | Predose and 0 to 72 hours postdose
  AUC (0-last) defined as the area under the analyte concentration-time curve from time zero to time of the last measurable (non-BQL) analyte concentration, calculated by linear-linear trapezoidal summation.
Plasma analyte concentration 24 hours (C24) Post Dose of Selexipag and ACT-333679 | Predose and 0 to 72 hours postdose
  C24 defined as plasma analyte concentration at 24 hours postdose.
Area Under the Analyte Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose and 0 to 72 hours postdose
  AUC (0-infinity) is defined the area under the analyte concentration-time curve from time zero to infinity time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable concentration, and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 50 Days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment and can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency